CLINICAL TRIAL: NCT01929382
Title: A Randomized, Double-Blind, Crossover Study to Determine the Effect of Actimmune® Dose Titration on the Severity and Incidence of Interferon Gamma-1b-Related Flu-Like Symptoms and the Pattern of Dropouts in Healthy Volunteers
Brief Title: Determining the Effect of Actimmune (Interferon Gamma 1b)Dose Titration on Flu-Like Symptoms in Healthy Volunteers
Acronym: FLS
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Vidara Therapeutics Research Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: VTRL Clin 2013-001
Record Dates: First submitted 2013-08-22; First posted 2013-08-27 (Estimated); Last update posted 2013-08-28 (Estimated); Status verified 2013-08

CONDITIONS: Adverse Effects in the Therapeutic Use of Interferon
Keywords: dose titration; FLS; flu like symptoms; Actimmune
MeSH Terms: interventions — Interferon-gamma; interferon gamma-1b

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Actimmune (interferon gamma 1b) (Active Comparator): Subjects > 0.5m2 BSA will receive 50 mcg/m2 BSA and subjects ≤ 0.5m2 BSA will receive 1.5mcg/kg/dose, as SC injections three times weekly, from week 1 to week 3.
  Interventions: Drug: interferon gamma 1b
- Actimmune(interferon gamma 1b) titration (Experimental): 30% of the recommended dose as SC injections three times weekly in week 1, 60% the recommended dose as SC injections three times weekly in week 2, and at the recommended dose as SC injections three times weekly in week 3
  Interventions: Drug: interferon gamma 1b

INTERVENTIONS:
Drug: interferon gamma 1b — Standard therapy vs dose titration
  Other Names: Actimmune

SUMMARY:
The most frequent side effects associated with Actimmune (interferon gamma 1b) therapy are the occurrence of 'flu-like symptoms' (FLS),which might include fever, chills, muscle aches, and tiredness. Earlier studies have demonstrated that these symptoms are common in healthy volunteers as well as in patients.

This study is designed to determine whether a titration of dosing reduces the frequency and severity of the FLS. A reported study with another interferon (interferon beta), demonstrated a reduction in the frequency and severity of the FLS when a titration of dosing was used. This study will compare the effects of the standard dose regimen with a titration regimen in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Ability to understand purpose & risks
* BMI 18-32kg/m2
* Females on contraception

Exclusion Criteria:

* History of HIV,or pos test for HCV Ab,or HBsAg
* History of chronic fatigue syndrome or fibromyalgia
* Flu like illness within 1 month of start
* History of depression or other mood disorder
* History of malignant or pre-malignant disease
* History of severe allergic reactions
* Known allergy to Actimmune or its components
* History of major diseases
* Clinically Significant abnormal labs
* Pregnant or breastfeeding
* Clinically abnormal ECG
* History of alcohol or substance abuse
* Other study participation in last 4 weeks
* Serious infection within 3 months
* Use of Rx products within 4 weeks except contraceptives or dermatology products
* Vaccinations within 2 weeks
* Tobacco products ( with limitations)
* Cant/wont comply with study requirements
* Allergy shots within 1 month
* Blood donation with limitations
* Investigator discretion as to unsuitability

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2013-07; Primary Completion 2013-09 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Change in severity of FLS vs baseline | 8 hrs post injection, thru 3 weeks of treatment

SECONDARY OUTCOMES:
Subject dropout rate | over 3 week study treatment

OTHER OUTCOMES:
Change in severity of FLS vs baseline | At 4 & 12 hours post injection

CONTACTS AND LOCATIONS:
Overall Officials: Mark Matson, MD, Principal Investigator — Prism Research Inc
Locations (1):
- Prism Research Inc, Saint Paul, Minnesota, United States

REFERENCES:
- [Background] Matson MA, Zimmerman TR Jr, Tuccillo D, Tang Y, Deykin A. Dose titration of intramuscular interferon beta-1a reduces the severity and incidence of flu-like symptoms during treatment initiation. Curr Med Res Opin. 2011 Dec;27(12):2271-8. doi: 10.1185/03007995.2011.630720. Epub 2011 Oct 28. PMID 21988668
- [Derived] Devane JG, Martin ML, Matson MA. A short 2 week dose titration regimen reduces the severity of flu-like symptoms with initial interferon gamma-1b treatment. Curr Med Res Opin. 2014 Jun;30(6):1179-87. doi: 10.1185/03007995.2014.899209. Epub 2014 Mar 13. PMID 24576196